CLINICAL TRIAL: NCT03372707
Title: Cuff Leak Test and Airway Obstruction in Mechanically Ventilated ICU Patients Pilot Trial
Brief Title: Cuff Leak Test and Airway Obstruction in Mechanically Ventilated ICU
Acronym: COMIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 20170701
Record Dates: First submitted 2017-12-01; First posted 2017-12-14 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Laryngeal Edema
Keywords: Cuff leak test; Post-extubation airway obstruction; Laryngeal edema
MeSH Terms: conditions — Laryngeal Edema

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients, Research Coordinators, study investigators, adjudicators, and data analysts will be blinded to the results of CLT in the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Patients randomized to the intervention arm will have the results of the Cuff Leak Test (CLT) (whether failed or passed) communicated to the treating physician; the treating physician will decide whether to proceed with extubation or not based on the CLT results. It is at the discretion of the treating physician to provide corticosteroids (4-5 mg of intravenous dexamethasone every six hours for up to 24 hours, with the last dose given one hour preceding extubation) and/or delay extubation by 24 hours should the patient fail the CLT.
  Interventions: Diagnostic Test: Cuff Leak Test
- Control Arm (No Intervention): In the control arm of this trial; the treating physicians and healthcare workers will be blinded to the results of the Cuff Leak Test (CLT); therefore, the Respiratory Therapist (RT) will proceed with extubation without delay or administering systemic steroid, regardless to the CLT results.

INTERVENTIONS:
Diagnostic Test: Cuff Leak Test — The Respiratory Therapist (RT) will perform the CLT on all enrolled patients. The patients will first be switched to volume assist-control (V-AC) with a respiratory rate of 10 breaths/min (to allow patient assist), constant flow of 60 l/min, and tidal volume set to match the average tidal volume currently being delivered during supportive ventilation. The RT will document the average exhaled volume over 3-5 breaths after switching to V-AC. The test will be performed by deflating the ETT balloon cuff with a 10 cc syringe, and: a) auscultation with a stethoscope to identify audible air leak around the ETT, and b) measuring the difference between the average exhaled volume prior to cuff deflation and the average exhaled volume over 3-5 breaths after cuff deflation.
  Arms: Intervention Arm

SUMMARY:
Introduction: Endotracheal intubation and mechanical ventilation are lifesaving interventions that are commonly done in the intensive care unit (ICU). The act of intubating someone can cause laryngeal edema (LE) that, if extensive enough, can cause airway obstruction after a patient is extubated. To date, the only test that is available to predict this complication is the cuff leak test (CLT). However, its diagnostic accuracy is uncertain as there have been no randomized controlled trials (RCT) examining this. The Cuff leak and airway Obstruction in Mechanically ventilated ICU patients (COMIC) Randomized Control Trial will be done to examine the impact of CLT on postextubation stridor and reintubation. Subsequently, describing the diagnostic accuracy of this test.

Methods: This will be a multi-center centered, pragmatic, double blinded RCT. Mechanically ventilated patients in the ICU, who are deemed ready to be extubated will be included. All patients will have a CLT done prior to extubation. The results of the CLT in the intervention arm will be communicated to the treating physician, and decision to extubate will be left to the treating team, while the results of the CLT for patients in the control arm will not be communicated to the treating physician, and the patient will be extubated, regardless of the result of the CLT.

Objective: This is a pilot trial to assess feasibility of conducting a powered RCT. Feasibility outcomes include: consent rate, recruitment rate, and protocol adherence. Clinical outcomes will include postextubation stridor, reintubation, emergency surgical airway, ICU mortality, in hospital mortality, duration of mechanical ventilation, and ICU length of stay in days.

DETAILED DESCRIPTION:
INTRODUCTION Endotracheal intubation and mechanical ventilation are lifesaving interventions. However, as with acute interventions, can be associated with serious complications. One such complication is laryngeal edema (LE) that occurs in 4-55% of patients. LE is thought to be caused by marked polymorphonuclear infiltration to the traumatized upper airway postintubation. The incidence of LE increases as the duration of intubation accrues, but it can occur as early as the first 24 hours of intubation. LE can result in airway narrowing and increased airflow velocity. It is postulated that narrowing of the lumen by 50% or more may result in postextubation stridor and respiratory distress. As a result, 3.5% (range 0-10.5%) of patients with LE will fail an extubation attempt and require reintubation. For various reasons, reintubation has a significant morbidity and mortality.

Identifying patients with LE can be challenging, the presence of the endotracheal tube (ETT) precludes direct visualization of the upper airway prior to extubation, therefore, clinicians cannot accurately predict airway obstruction before it occurs. A cuff-leak test (CLT) was first described in 1988 as a surrogate for direct visualization and a screening for airway edema prior to extubation. This test involves deflating the balloon cuff on an ETT and observing if the patient is able to breathe around it. If air can pass around the ETT, it suggest that the airway is patent and clinicians may proceed with extubation. A small leak or complete absence of one, would suggest an airway obstruction.

There are conflicting results on the utility and accuracy of a CLT. To date, two meta-analyses of observational studies examined the diagnostic accuracy of a CLT. One meta-analysis reports that a failed CLT is insensitive but a specific predictor of LE (pooled sensitivity and specificity 0.56; 95% CI, 0.48-0.63 and 0.92; 95% CI, 0.90-0.93, respectively) and reintubation (pooled sensitivity and specificity for reintubation 0.63; 95% CI, 0.38-0.84 and 0.86; 95% CI, 0.81-0.90, respectively). While the second meta-analysis also states that the failed CLT was associated with postextubation LE, particularly in patients with > 5 days duration of intubation (odds ratio [OR]=2.09; 95% CI, 1.28-2.89), it was not associated with higher odds of reintubation (OR=0.94; 95% CI, 0.32-1.57).

Despite the lack of high quality studies, an absent cuff leak usually results in delayed extubation and exposure to corticosteroids to empirically treat airway edema. A recent meta-analysis of 11 parallel randomized controlled trails (RCTs) with a total of 2472 patients examined the effect of prophylactic corticosteroids prior to extubation on postextubation stridor and reintubation. Prophylactic corticosteroids use reduced the risk of postextubation airway events when compared to placebo or no treatment (RR 0.43; 95% CI 0.29-0.66, P=0.002). A subgroup analysis demonstrates that this benefit is only significant in patients that are deemed "high risk" for LE. Prophylactically treating unspecified patients shows no reduction in postextubation events and exposes patients to high dose steroids (16). Moreover, a false positive CLT can unnecessarily delay extubation, leading to a prolonged length of stay in the intensive care unit (ICU), barotraumas, and increased risk of ventilator associated pneumonias, therefore, exposing patients unnecessarily to these undesirable outcomes. On the other hand, if a CLT is not performed, or if in case of a false negative test, some patients may fail the extubation attempt and require reintubation.

Recent clinical practice guidelines for using CLT reflect this uncertainty. The American Thoracic Society guidelines on liberation of mechanical ventilation issued a weak recommendation for performing CLT in mechanically ventilated adults who are at high risk for postextubation stridor (conditional recommendation, very low certainty). There is also significant clinical equipoise. A recent unpublished survey found that 42% (12/26) of Canadian intensive care unit (ICU) physicians either never or rarely request to know the results of a cuff leak test prior to extubating a patient that is at moderate risk of laryngeal edema while 23% will always or usually order the test. Therefore, a large RCT is necessary to investigate the diagnostic accuracy of the CLT and its impact on patients' outcomes.

Herein, the investigators are reporting the protocol for the COMIC Pilot Trial. The COMIC (Cuff leak and airway Obstruction in Mechanically ventilated ICU patients) pilot trial will be a multicenter, randomized, concealed, blinded, parallel-group, pragmatic pilot trial. The purpose is to determine the feasibility of undertaking a powered RCT to examine the impact of CLT on postextubation stridor and reintubation. Subsequently, describing the diagnostic accuracy of this test.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be mechanically ventilated adults (>18 years) who are admitted to the ICU and an order to extubate has been provided by the treating physician.

Exclusion Criteria:

1. A palliative care, a one-way extubation, or a decision to withdraw advances life support order has been written.
2. Pregnancy.
3. Patients at high risk for LE: burn patients, smoke inhalation injuries (as defined as singed facial hair or nasal hair, carbonaceous secretions/sputum, and known to be in an enclosed fire), blunt or penetrating trauma involving the neck and airway, postoperative head and neck surgeries, and patients admitted with airway edema to the ICU (e.g; anaphylaxis).
4. Patients with either a difficult or traumatic endotracheal intubation.
5. Patients receiving mechanical ventilation via tracheostomy.
6. Known preexisting tracheolaryngeal abnormalities such as: vocal cord paralysis, tracheolaryngeal neoplasm, tracheomalacia, tracheolaryngeal stenosis, or previous head and neck surgeries.
7. Patients receiving systemic corticosteroids of greater than 30 mg of PO prednisone or equivalent, within 4 days prior to the decision to extubate.
8. Patients who failed extubation attempt within the current ICU admission.
9. History of postextubation airway obstruction.
10. The ICU physician declined enrolling the patient.
11. Patient had a failed CLT in the previous 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Consent Rate | 1 year
  A successful consent rate will be defined as 70% of substitute decision makers (SDMs) or patients approached to consent, choosing to participate in the trial. This will be calculated as the overall proportion of SDMs or patients consenting out of those approached (with 95% CI). Note that a mixed consent model will be obtained. In Canada and Saudi Arabia, a priori or deferred consent model will be used. In Poland, a waved consent model will be used.
Recruitment Rate | 1 year
  A successful recruitment rate will be defined as achieving enrollment of 40 patients, conventionally expressed as four patients per month over the duration of the trial. While the pilot trial is ongoing, recruitment will be reviewed weekly and the screening records will be reviewed monthly with the cases of missed eligible patients reviewed. If applicable, barriers to enrollment will be addressed to maximize recruitment. The recruitment metric will be measured and interpreted at the end of the pilot trial by calculating the mean number of recruited patients per active screening month.
Protocol Adherence | 1 year
  Successful adherence will be defined as ≥80%. The adherence will be calculated as the proportion of patients that were assigned to the control arm being extubated after CLT being performed and the portion of people that assigned to the intervention arm who are given the prescribed steroids for a failed CLT. As this pilot trial is ongoing, investigators will review adherence monthly and investigate the reasons for compliance failure. All reasons for either failure to extubate after a failed CLT in the control arm will be investigated. The RC will review the Respiratory Therapists' notes, and the medication profile to determine actual compliance. All reasons for non-compliance will be recorded for both groups using distinguishing clinical reasons (eg. Palliation, death, consent withdrawal, errors).

SECONDARY OUTCOMES:
Postextubation stridor | 48 hours after original extubation
  Defined as an audible high pitched inspiratory noise caused by turbulent airflow through the narrowed airway that is detectable with or without a stethoscope within 48 hours of extubation.
Clinically significant postextubation stridor | 48 hours after original extubation
  Defined as stridor (see definition above) that requires medical intervention such as the administration of systemic steroids, racemic epinephrine, or Heli-ox.
Reintubation | 72 hours after original extubation
  Defined as reintubation within 72 hours of original extubation while in the ICU.
Emergency surgical airway | 30 days
  Defined as performing urgent tracheotomy or cricothyroidotomy for a life-threatening airway obstruction
In ICU mortality | 1 year
In hospital mortality truncated at 30 days | 30 days
Duration of mechanical ventilation | 1 year
  Defined as time on the ventilator after randomization in days.
ICU length of stay in days | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kimberley A Lewis, MD, Principal Investigator — McMaster University; Waleed Alhazzani, MD, Principal Investigator — McMaster University
Locations (3):
- St Joseph's Hospital, Hamilton, Ontartio, Canada
- Jagiellonian University Medical College, Krakow, Lesser Poland Voivodeship, Poland
- Imam Adbulrahman Bin Faisal University, Dammam, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maury E, Guglielminotti J, Alzieu M, Qureshi T, Guidet B, Offenstadt G. How to identify patients with no risk for postextubation stridor? J Crit Care. 2004 Mar;19(1):23-8. doi: 10.1016/j.jcrc.2004.02.005. PMID 15101002
- [Background] Tadie JM, Behm E, Lecuyer L, Benhmamed R, Hans S, Brasnu D, Diehl JL, Fagon JY, Guerot E. Post-intubation laryngeal injuries and extubation failure: a fiberoptic endoscopic study. Intensive Care Med. 2010 Jun;36(6):991-8. doi: 10.1007/s00134-010-1847-z. Epub 2010 Mar 18. PMID 20237758
- [Background] Sutherasan Y, Theerawit P, Hongphanut T, Kiatboonsri C, Kiatboonsri S. Predicting laryngeal edema in intubated patients by portable intensive care unit ultrasound. J Crit Care. 2013 Oct;28(5):675-80. doi: 10.1016/j.jcrc.2013.05.011. Epub 2013 Jun 24. PMID 23806246
- [Background] Francois B, Bellissant E, Gissot V, Desachy A, Normand S, Boulain T, Brenet O, Preux PM, Vignon P; Association des Reanimateurs du Centre-Ouest (ARCO). 12-h pretreatment with methylprednisolone versus placebo for prevention of postextubation laryngeal oedema: a randomised double-blind trial. Lancet. 2007 Mar 31;369(9567):1083-9. doi: 10.1016/S0140-6736(07)60526-1. PMID 17398307
- [Background] Zhou T, Zhang HP, Chen WW, Xiong ZY, Fan T, Fu JJ, Wang L, Wang G. Cuff-leak test for predicting postextubation airway complications: a systematic review. J Evid Based Med. 2011 Nov;4(4):242-54. doi: 10.1111/j.1756-5391.2011.01160.x. PMID 23672755
- [Background] Way WL, Sooy FA. Histologic changes produced by endotracheal intubation. Ann Otol Rhinol Laryngol. 1965 Sep;74(3):799-812. doi: 10.1177/000348946507400318. No abstract available. PMID 4954421
- [Background] Mackle T, Meaney J, Timon C. Tracheoesophageal compression associated with substernal goitre. Correlation of symptoms with cross-sectional imaging findings. J Laryngol Otol. 2007 Apr;121(4):358-61. doi: 10.1017/S0022215106004142. Epub 2006 Oct 26. PMID 17064460
- [Background] Epstein SK, Ciubotaru RL. Independent effects of etiology of failure and time to reintubation on outcome for patients failing extubation. Am J Respir Crit Care Med. 1998 Aug;158(2):489-93. doi: 10.1164/ajrccm.158.2.9711045. PMID 9700126
- [Background] Demling RH, Read T, Lind LJ, Flanagan HL. Incidence and morbidity of extubation failure in surgical intensive care patients. Crit Care Med. 1988 Jun;16(6):573-7. doi: 10.1097/00003246-198806000-00001. PMID 3371019
- [Background] Esteban A, Alia I, Gordo F, Fernandez R, Solsona JF, Vallverdu I, Macias S, Allegue JM, Blanco J, Carriedo D, Leon M, de la Cal MA, Taboada F, Gonzalez de Velasco J, Palazon E, Carrizosa F, Tomas R, Suarez J, Goldwasser RS. Extubation outcome after spontaneous breathing trials with T-tube or pressure support ventilation. The Spanish Lung Failure Collaborative Group. Am J Respir Crit Care Med. 1997 Aug;156(2 Pt 1):459-65. doi: 10.1164/ajrccm.156.2.9610109. PMID 9279224
- [Background] Frutos-Vivar F, Esteban A, Apezteguia C, Gonzalez M, Arabi Y, Restrepo MI, Gordo F, Santos C, Alhashemi JA, Perez F, Penuelas O, Anzueto A. Outcome of reintubated patients after scheduled extubation. J Crit Care. 2011 Oct;26(5):502-509. doi: 10.1016/j.jcrc.2010.12.015. Epub 2011 Mar 3. PMID 21376523
- [Background] Torres A, Gatell JM, Aznar E, el-Ebiary M, Puig de la Bellacasa J, Gonzalez J, Ferrer M, Rodriguez-Roisin R. Re-intubation increases the risk of nosocomial pneumonia in patients needing mechanical ventilation. Am J Respir Crit Care Med. 1995 Jul;152(1):137-41. doi: 10.1164/ajrccm.152.1.7599812.
- [Background] Seymour CW, Martinez A, Christie JD, Fuchs BD. The outcome of extubation failure in a community hospital intensive care unit: a cohort study. Crit Care. 2004 Oct;8(5):R322-7. doi: 10.1186/cc2913. Epub 2004 Jul 20. PMID 15469575
- [Background] Potgieter PD, Hammond JM. "Cuff" test for safe extubation following laryngeal edema. Crit Care Med. 1988 Aug;16(8):818. doi: 10.1097/00003246-198808000-00020. No abstract available. PMID 3396380
- [Background] Ochoa ME, Marin Mdel C, Frutos-Vivar F, Gordo F, Latour-Perez J, Calvo E, Esteban A. Cuff-leak test for the diagnosis of upper airway obstruction in adults: a systematic review and meta-analysis. Intensive Care Med. 2009 Jul;35(7):1171-9. doi: 10.1007/s00134-009-1501-9. Epub 2009 Apr 28. PMID 19399474
- [Background] Kuriyama A, Umakoshi N, Sun R. Prophylactic Corticosteroids for Prevention of Postextubation Stridor and Reintubation in Adults: A Systematic Review and Meta-analysis. Chest. 2017 May;151(5):1002-1010. doi: 10.1016/j.chest.2017.02.017. Epub 2017 Feb 21. PMID 28232056
- [Background] Girard TD, Alhazzani W, Kress JP, Ouellette DR, Schmidt GA, Truwit JD, Burns SM, Epstein SK, Esteban A, Fan E, Ferrer M, Fraser GL, Gong MN, Hough CL, Mehta S, Nanchal R, Patel S, Pawlik AJ, Schweickert WD, Sessler CN, Strom T, Wilson KC, Morris PE; ATS/CHEST Ad Hoc Committee on Liberation from Mechanical Ventilation in Adults. An Official American Thoracic Society/American College of Chest Physicians Clinical Practice Guideline: Liberation from Mechanical Ventilation in Critically Ill Adults. Rehabilitation Protocols, Ventilator Liberation Protocols, and Cuff Leak Tests. Am J Respir Crit Care Med. 2017 Jan 1;195(1):120-133. doi: 10.1164/rccm.201610-2075ST. PMID 27762595
- [Background] Altinok T, Can A. Management of tracheobronchial injuries. Eurasian J Med. 2014 Oct;46(3):209-15. doi: 10.5152/eajm.2014.42. Epub 2014 Aug 26. PMID 25610327
- [Background] Law JA, Broemling N, Cooper RM, Drolet P, Duggan LV, Griesdale DE, Hung OR, Jones PM, Kovacs G, Massey S, Morris IR, Mullen T, Murphy MF, Preston R, Naik VN, Scott J, Stacey S, Turkstra TP, Wong DT; Canadian Airway Focus Group. The difficult airway with recommendations for management--part 1--difficult tracheal intubation encountered in an unconscious/induced patient. Can J Anaesth. 2013 Nov;60(11):1089-118. doi: 10.1007/s12630-013-0019-3. Epub 2013 Oct 17. PMID 24132407
- [Background] Smith OM, McDonald E, Zytaruk N, Foster D, Matte A, Clarke F, Fleury S, Krause K, McArdle T, Skrobik Y, Cook DJ. Enhancing the informed consent process for critical care research: strategies from a thromboprophylaxis trial. Intensive Crit Care Nurs. 2013 Dec;29(6):300-9. doi: 10.1016/j.iccn.2013.04.006. Epub 2013 Jul 18. PMID 23871290
- [Background] Alhazzani W, Guyatt G, Alshahrani M, Deane AM, Marshall JC, Hall R, Muscedere J, English SW, Lauzier F, Thabane L, Arabi YM, Karachi T, Rochwerg B, Finfer S, Daneman N, Alshamsi F, Zytaruk N, Heel-Ansdell D, Cook D; Canadian Critical Care Trials Group. Withholding Pantoprazole for Stress Ulcer Prophylaxis in Critically Ill Patients: A Pilot Randomized Clinical Trial and Meta-Analysis. Crit Care Med. 2017 Jul;45(7):1121-1129. doi: 10.1097/CCM.0000000000002461. PMID 28459708
- [Background] Ouellette DR, Patel S, Girard TD, Morris PE, Schmidt GA, Truwit JD, Alhazzani W, Burns SM, Epstein SK, Esteban A, Fan E, Ferrer M, Fraser GL, Gong MN, Hough CL, Mehta S, Nanchal R, Pawlik AJ, Schweickert WD, Sessler CN, Strom T, Kress JP. Liberation From Mechanical Ventilation in Critically Ill Adults: An Official American College of Chest Physicians/American Thoracic Society Clinical Practice Guideline: Inspiratory Pressure Augmentation During Spontaneous Breathing Trials, Protocols Minimizing Sedation, and Noninvasive Ventilation Immediately After Extubation. Chest. 2017 Jan;151(1):166-180. doi: 10.1016/j.chest.2016.10.036. Epub 2016 Nov 3. PMID 27818331
- [Derived] Lewis K, Culgin S, Jaeschke R, Perri D, Marchildon C, Hassall K, Almubarak Y, Szczeklik W, Piraino T, Thabane L, Alqahtani KM, Alghamdi A, Alshahrani M, Alhazzani W. Cuff Leak Test and Airway Obstruction in Mechanically Ventilated Intensive Care Unit Patients: A Pilot Randomized Controlled Clinical Trial. Ann Am Thorac Soc. 2022 Feb;19(2):238-244. doi: 10.1513/AnnalsATS.202103-390OC. PMID 34242140
- [Derived] Lewis K, Culgin S, Jaeschke R, Perri D, Marchildon C, Hassall K, Piraino T, Thabane L, Almubarak Y, Alshahrani MS, Rochwerg B, Baw B, Szczeklik W, Karachi T, Alhazzani W; GUIDE Group. Cuff Leak Test and Airway Obstruction in Mechanically Ventilated ICU Patients (COMIC): a pilot randomised controlled trial protocol. BMJ Open. 2019 Jul 19;9(7):e029394. doi: 10.1136/bmjopen-2019-029394. PMID 31326936

DOCUMENTS (1):
  • Study Protocol (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT03372707/Prot_000.pdf